CLINICAL TRIAL: NCT05943574
Title: Post-Market Clinical Follow-Up Study to Provide Safety, Performance and Clinical Benefits Data of the XtraFix® Small External Fixation System (Implants and Instrumentation) - A Retrospective Consecutive Series Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the XtraFix® Small External Fixation System
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-147T
Record Dates: First submitted 2023-05-22; First posted 2023-07-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Wrist Fracture; Proximal Humerus Fracture
Keywords: Post-Market Clinical Follow-Up Study; Medical Device; Performance; Clinical Benefits; Safety; Wrist Fracture; Humerus Fracture
MeSH Terms: conditions — Wrist Fractures; Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received the XtraFix® Small External Fixation System

SUMMARY:
The study is a monocentric, retrospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to confirm safety, performance and clinical benefits of the XtraFix® Small External Fixation System (implants and instrumentation) when used to treat long bone fractures.

The primary objective is the assessment of performance by analyzing fracture healing.

The secondary objectives are the assessment of safety by recording and analyzing the incidence and frequency of complications and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified. Subjects' outcomes will also be assessed.

DETAILED DESCRIPTION:
The XtraFix® Small External Fixation System is intended to be used for the treatment of appropriately sized long bone fractures (in foot, arm, wrist and hand), which account for 20% of all fractures in emergency departments and are the most common fractures in all patients under the age of 75. In this study we will only collect data on wrist and proximal humerus fractures.

One site will be involved in this study. The aim is to include a maximum of 91 consecutive series cases who received the XtraFix® Small External Fixation System at the Azienda Ospedaliera di Rilievo Nazionale "Antonio Cardarelli" (Naples, Italy) starting from 2019 until 2021. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preoperative, intraoperative, immediate post-operative and device removal visit will be available in medical notes and collected retrospectively. During a follow up phone call at least 1 year post-operative the subject will be asked to complete a patient questionnaire and a clinical assessment of the fracture healing will be done. In addition, any complications since the last consultation visit at the clinic and information about the treatment of the complications will also be collected over the phone.

ELIGIBILITY:
Inclusion Criteria:

* 18-year-old or older patients having received the XtraFix® Small External Fixation System for the treatment of long bone fractures.
* Specifically, the system is intended for temporary stabilization of open or closed fractures, typically in the context of polytrauma or where open or alternative closed treatment is undesirable or otherwise contraindicated.
* Revision surgeries will also be included in the study.
* In this study we will only collect data on wrist and proximal humerus fractures.

Exclusion Criteria:

* Off-label use
* Active or suspected infection
* Conditions that limit the patient's ability and/or willingness to follow instructions during the healing process
* Inadequate skin, bone, or neurovascular status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of cases implanted with the XtraFix® Small External Fixation System according to Zimmer Biomet's Instruction for Use (IFU) and who meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Performance: Fracture healing assessed radiographically or clinically. | Radiographically at the Device Removal Visit up to 1 year postoperative or clinically at the Follow-Up Phone call at least 1 year postoperative.
  When radiographs are not available, the fracture healing will be assessed clinically (pain at fracture site).

SECONDARY OUTCOMES:
Product safety will be assessed by recording the complications and adverse events. | At time of the surgery, immediate post-operative, at the Device Removal Visit up to 1 year postoperative and at the Follow-Up Phone Call at least 1 year postoperative.
  Incidence and frequency of complications and adverse events will be assessed by recording them any time they occur until the Follow-up phone call at minimum 1 year postoperative.
EuroQol five-dimensional Health Questionnaire (EQ-5D-5L) | At the Follow-Up Phone Call at least 1 year postoperative.
  Assessment of patient-reported outcome measures (PROMs): The EuroQol fivedimensional Health Questionnaire (EQ-5D-5L) is a generic instrument. The EQ-5D-5L is scored on a 0 to 100 mm scale. 0 mm represents "the worst..." and 100 mm represents "the best health you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- Azienda Ospedaliera di Rilievo Nazionale "Antonio Cardarelli", Naples, Campania, Italy